CLINICAL TRIAL: NCT01961869
Title: Phytochemical Release Rate From Black Raspberry Confections Alters Gene Expression and Chemical Profiles Relevant to Inhibition of Oral Carcinogenesis
Brief Title: Black Raspberry Confection in Preventing Oral Cancer in Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Yael Vodovotz, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-13052; NCI-2013-01724 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers
Keywords: black raspberry; chemoprevention; oral delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm I (Fast release BRB confection 4g) (Experimental): Participants receive one fast release BRB confection (4g) PO 4-6 hours apart thrice daily (TID) for 2 weeks.
  Interventions: Other: Fast release BRB confection
- Arm II (Fast release BRB confection 8g) (Experimental): Participants receive two fast release BRB confection (8g) PO 4-6 hours apart TID for 2 weeks.
  Interventions: Other: Fast release BRB confection
- Arm III (Intermed release BRBconfection 4g) (Experimental): Participants receive one intermediate release BRB confection (4g) PO 4-6 hours apart TID for 2 weeks.
  Interventions: Other: Intermed release BRB confection
- Arm IV (Intermed release BRBconfection 8g) (Experimental): Participants receive two intermediate release BRB confection (8g) PO 4-6 hours apart TID for 2 weeks.
  Interventions: Other: Intermed release BRB confection
- Arm V (Prolong release BRB confection 4g) (Experimental): Participants receive one prolonged release BRB confection (4g) PO 4-6 hours apart TID for 2 weeks.
  Interventions: Other: Prolong release BRB confection
- Arm VI (Prolong release BRB confection 8g) (Experimental): Participants receive two prolonged release BRB confection (8g) PO 4-6 hours apart TID for 2 weeks.
  Interventions: Other: Prolong release BRB confection

INTERVENTIONS:
Other: Fast release BRB confection — Fast release BRB confection includes lyophilized black raspberry powder, corn syrup, and sugar. All ingredients are generally regarded as safe (GRAS) food ingredients
  Other Names: black raspberry confection; BRB confection; LBR lozenge
  Arms: Arm I (Fast release BRB confection 4g); Arm II (Fast release BRB confection 8g)
Other: Intermed release BRB confection — Intermediate release BRB confection includes lyophilized black raspberry powder, corn syrup, sugar, and pectin. All ingredients are generally regarded as safe (GRAS) food ingredients
  Other Names: black raspberry confection; BRB confection; LBR lozenge
  Arms: Arm III (Intermed release BRBconfection 4g); Arm IV (Intermed release BRBconfection 8g)
Other: Prolong release BRB confection — Prolonged release BRB confection includes lyophilized black raspberry powder, corn syrup, corn starch, and sugar. All ingredients are generally regarded as safe (GRAS) food ingredients.
  Other Names: black raspberry confection; BRB confection; LBR lozenge
  Arms: Arm V (Prolong release BRB confection 4g); Arm VI (Prolong release BRB confection 8g)

SUMMARY:
This clinical trial studies black raspberry confection in preventing oral cancer in healthy volunteers. Black raspberry contains ingredients that may prevent or slow the growth of certain cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To select an optimal black raspberry confection based on altered gene expression and chemical profiles in healthy individuals exposed to 3 black raspberry-based amorphous functional confections with modulated bioactive release rate at two doses (4 g and 8 g).

OUTLINE: Participants are randomized to 1 of 6 arms after 2 weeks.

ARM I: Participants receive black raspberry (BRB) confection 1 fast release orally (PO) 4-6 hours apart thrice daily (TID) for 2 weeks.

ARM II: Participants receive BRB confection 2 fast release PO 4-6 hours apart TID for 2 weeks.

ARM III: Participants receive BRB confection 1 intermediate release PO 4-6 hours apart TID for 2 weeks.

ARM IV: Participants receive BRB confection 2 intermediate release PO 4-6 hours apart TID for 2 weeks.

ARM V: Participants receive BRB confection 1 prolonged release PO 4-6 hours apart TID for 2 weeks.

ARM VI: Participants receive BRB confection 2 prolonged release PO 4-6 hours apart TID for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy, free-living adults
* Be a non-smoker (defined as adults who have never smoked or who have not had a cigarette in the past ten years)
* Agree to consume a standardized vitamin/mineral supplement and avoid other nutrition and alternative supplements for the duration of the study
* Agree to follow a berry-restricted diet and to document any accidental consumption of restricted foods each day of the study
* Agree to abstain from mouthwashes

Exclusion Criteria:

* Have an active metabolic or digestive illness including malabsorptive disorders, renal insufficiency, hepatic insufficiency, cachexia, or short bowel syndrome
* Have an active or a recent history of any condition that causes altered immunity such as chronic inflammatory disease, autoimmune disorders, cancer, anemia, and blood dyscrasias
* Have a known allergy or food intolerance to ingredients in study products (black raspberries),other berries, wheat, or soy
* Are strict vegans (no consumption of animal, fish or egg products)
* Are planning to conceive, or are currently pregnant or lactating
* Are heavy alcohol consumers (defined as an average consumption of greater than 2 drinks/day)
* Have a history of oral cancer or currently undergoing treatment of oral cancer
* In the last month have had any active oral lesions or maladies or currently have any oral disease or obvious open sores in the oral cavity or surrounding the oral opening
* Have strong gag reflex or problems swallowing that prohibit buccal brushing of the oral cavity
* Have been on an antibiotic regime lasting for one week in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2014-05-14 (Actual); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Acceptance of candidate formulations, assessed using a 9 point hedonic scale (1 =dislike very much, 9 = like very much) | Up to day 14
  Compliance and safety of the confections will be evaluated using dietary and sensory questionnaires. The analysis of variance (ANOVA) style model accounting for the random effect of the individual subject and the fixed effect of the dissolution (amorphous confection form) group will be used to examine the effect of attribute data, gender, and age using a 9-point hedonic scale. The significant differences between means of the different groups will be examined using the Ryan-Einot-Gabriel-Welsch (REGW) multiple comparisons test.
Bioavailability index, defined as the average rank of BRB effect in anthocyanins, ellagic acid, urolithins, and quercetin derivatives | Up to day 14
  To select an optimal delivery vehicle & dose, a combination that results in any of 10 subjects having an adverse event will be eliminated in the 1st stage. In the 2nd and 3rd stages ANOVA style models accounting for the random effect of individual subject and the fixed effect of dose & release rate will be used to examine phytonutrient metabolite & gene expression. Using the multiple comparisons with the best procedure, any combination will be eliminated that is significantly worse than the best combination for a global index of bioavailability (stage 2) and gene expression effects (stage 3).
Gene expression index, defined as the average rank of BRB effect on expression of genes responsive to BRBs and important to smoking and inflammatory response | Up to day 14
  To select an optimal delivery vehicle & dose, a combination that results in any of 10 subjects having an adverse event will be eliminated in the 1st stage. In the 2nd and 3rd stages ANOVA style models accounting for the random effect of individual subject and the fixed effect of dose & release rate will be used to examine phytonutrient metabolite & gene expression. Using the multiple comparisons with the best procedure, any combination will be eliminated that is significantly worse than the best combination for a global index of bioavailability (stage 2) and gene expression effects (stage 3).

CONTACTS AND LOCATIONS:
Overall Officials: Yael Vodovotz, Ph.D., Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu